CLINICAL TRIAL: NCT04776148
Title: A Phase 3 Randomized Study of Lenvatinib in Combination With Pembrolizumab Versus Standard of Care in Participants With Metastatic Colorectal Cancer Who Have Received and Progressed On or After or Became Intolerant to Prior Treatment
Brief Title: Study of Lenvatinib (MK-7902/E7080) in Combination With Pembrolizumab (MK-3475) Versus Standard of Care in Participants With Metastatic Colorectal Cancer (MK-7902-017/E7080-G000-325/LEAP-017)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7902-017; MK-7902-017 (Other: MSD); LEAP-017 (Other: MSD); E7080-G000-325 (Other: Eisai); jRCT2031200453 (Registry Identifier: jRCT); 2020-004289-20 (EudraCT Number)
Record Dates: First submitted 2021-02-26; First posted 2021-03-01 (Actual); Results first posted 2024-04-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Neoplasms
Keywords: Programmed Cell Death Receptor 1 (PD-1); Programmed Cell Death Receptor Ligand 1 (PD-L1); Programmed Cell Death Receptor Ligand 2 (PD-L2); PD-1; PDL1; PD-L1; PD-L2
MeSH Terms: conditions — Colorectal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib; regorafenib; trifluridine tipiracil drug combination; Trifluridine; tipiracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- lenvatinib+pembrolizumab (Experimental): Participants receive pembrolizumab 400 mg via intravenous (IV) infusion on Day 1 of each 6-week (Q6W) Cycle for up to 18 cycles (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule once daily until progressive disease.
  Interventions: Drug: pembrolizumab; Drug: lenvatinib
- standard of care treatment (regorafenib OR TAS-102) (Active Comparator): Participants receive regorafenib 160 mg via oral tablet once daily on Days 1 through 21 of each 4-week cycle OR TAS-102 (trifluridine and tipiracil hydrochloride) 35 mg/m^2 via oral tablet twice a day on Days 1 through 5 and Days 8-12 of each 4-week cycle until progressive disease.
  Interventions: Drug: regorafenib; Drug: TAS-102 (trifluridine and tipiracil)

INTERVENTIONS:
Drug: pembrolizumab — IV infusion
  Other Names: KEYTRUDA®; MK-3475
  Arms: lenvatinib+pembrolizumab
Drug: lenvatinib — oral capsule
  Other Names: MK-7902; E7080
  Arms: lenvatinib+pembrolizumab
Drug: regorafenib — oral tablet
  Other Names: STIVARGA®; REGONIX®
  Arms: standard of care treatment (regorafenib OR TAS-102)
Drug: TAS-102 (trifluridine and tipiracil) — oral tablet
  Other Names: LONSURF®
  Arms: standard of care treatment (regorafenib OR TAS-102)

SUMMARY:
The purpose of this study is to assess the safety and efficacy of lenvatinib (MK-7902/E7080) in combination with pembrolizumab (MK-3475) in participants with metastatic colorectal cancer. The study will also compare lenvatinib plus pembrolizumab with the standard of care treatment of regorafenib and TAS-102 (trifluridine and tipiracil hydrochloride).

The primary study hypothesis is that lenvatinib plus pembrolizumab is superior to standard of care with respect to overall survival.

DETAILED DESCRIPTION:
The Global portion, or Global Cohort, will include all participants who are enrolled during the Global enrollment period and will be the primary analysis population for the study. After enrollment of the global portion of the study is complete, the study will remain open to enrollment in China alone until the target number of participants from China have been enrolled to meet local regulatory requirements.

The China Cohort will include both participants enrolled in China for the Global Cohort plus those participants enrolled in China as part of the China extension enrollment period.

Per the supplemental Statistical Analysis Plan (sSAP), China participants randomized after the enrollment of the global portion is closed as part of the China extension enrollment period will not be included in the global analysis populations.

As pre-specified in the protocol, safety and efficacy outcome measures for the China Cohort will be analyzed separately from the Global Cohort.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed diagnosis of unresectable and metastatic colorectal adenocarcinoma (Stage IV A, B and C as defined by American Joint Committee on Cancer [AJCC] 8th edition). Note: Tumor must be determined to be NOT microsatellite instability-high (MSI-H)/mismatch repair deficient (dMMR) by local testing
* Has been previously treated for their disease and has shown disease progression as defined by RECIST 1.1 on or after or could not tolerate standard treatment, which must include ALL of the following agents if approved and locally available in the country where the participant is randomized:

  1. fluoropyrimidine, irinotecan and oxaliplatin
  2. with or without an anti-vascular endothelial growth factor (VEGF) monoclonal antibody (bevacizumab)
  3. with anti- epidermal growth factor receptor (EGFR) monoclonal antibodies (cetuximab or panitumumab) for RAS (KRAS/NRAS) wild-type (WT) participants
  4. BRAF inhibitor (in combination with cetuximab +/- binimetinib) for BRAF V600E mutated metastatic colon cancer (mCRC)
* Has measurable disease per RECIST 1.1 assessed by the investigator
* Has provided to a designated central laboratory an archival tumor tissue sample or newly obtained core, incisional, or excisional biopsy of a tumor lesion which has not been previously irradiated
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 3 days prior to randomization
* Has a life expectancy of at least 3 months, based on the investigator assessment
* Has the ability to swallow capsules or ingest a suspension orally or by a feeding tube
* Has adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 millimeter of mercury (mmHg) with no change in antihypertensive medications within 1 week prior to randomization
* Male participants must agree to the following during the treatment period and for at least 90 days after the last dose of regorafenib or TAS-102 and at least 7 days after the last dose of lenvatinib: refrain from donating sperm PLUS either be abstinent from heterosexual intercourse as their preferred and usual lifestyle or use contraception. The male contraception period should continue for at least 7 days after discontinuation of lenvatinib
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: is not a woman of childbearing potential (WOCBP) OR is a WOCBP and using a highly-effective contraceptive method during the treatment period and for at least 30 days after the last dose of lenvatinib, 120 days after the last dose of pembrolizumab, and 180 days after the last dose of regorafenib or TAS-102 (whichever is last) AND agrees not to donate eggs (ova, oocytes)
* A WOCBP must have a negative highly sensitive pregnancy test (urine or serum) within 24 hours before the first dose of study treatment

Exclusion Criteria:

* Has a tumor that is microsatellite instability-high (MSI-H)/mismatch repair deficient (dMMR) per local testing
* Has presence of gastrointestinal condition, eg, malabsorption, that might affect the absorption of study drug.
* Has present or progressive accumulation of pleural, ascitic, or pericardial fluid requiring drainage or diuretic drugs within 2 weeks prior to enrollment
* Has radiographic evidence of encasement or invasion of a major blood vessel invasion or of intratumoral cavitation. In the chest, major blood vessels include the main pulmonary artery, the left and right pulmonary arteries, the 4 major pulmonary veins, the superior or inferior vena cava, and the aorta
* Has clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study drug
* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability.

Participants with cardiac failure NYHA Class II, III and IV are not allowed to be assigned to the regorafenib in Arm B

* Has a history of arterial thromboembolism within 12 months of start of study drug
* Has urine protein ≥1 gram/24 hour
* Has prolongation of QT interval corrected with Fridericia's formula (QTcF interval) to >480 milliseconds
* Has left ventricular ejection fraction (LVEF) below the institutional (or local laboratory) normal range as determined by multigated acquisition (MUGA) or echocardiogram (ECHO)
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years with certain exceptions
* Has serious nonhealing wound, ulcer or bone fracture
* Has had major surgery within 3 weeks prior to first dose of study treatment
* Has received biologic response modifiers (eg, granulocyte colony-stimulating factor) within 4 weeks before study entry
* Has preexisting ≥Grade 3 gastrointestinal or nongastrointestinal fistula
* Has received prior treatment with a combination of an anti-PD-1, anti-PD-L1, or anti PD-L2 agent with anti-VEGF monoclonal antibodies or vascular endothelial growth factor receptor (VEGFR) inhibitors
* Has previously received regorafenib or TAS-102
* Has received prior systemic anti-cancer therapy including investigational agents within 28 days prior to randomization
* Has received prior radiotherapy within 2 weeks of start of study treatment
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study treatment
* Has known intolerance to lenvatinib, regorafenib, or TAS-102 and/or any of their excipients
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 28 days prior to the first dose of study treatment
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of Human Immunodeficiency Virus (HIV) infection
* Has a known history of Hepatitis B or known active Hepatitis C virus infection
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (95):
- United States (12):
  - Pacific Cancer Care ( Site 0031), Monterey, California
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital ( Site 0021), Marietta, Georgia
  - University of Chicago Medical Center-Medicine - Section of Hematology/Oncology - Gastrointestinal P, Chicago, Illinois
  - MFSMC-HJWCI-Oncology Research ( Site 0012), Baltimore, Maryland
  - MedStar Good Samaritan Hospital-Oncology Research ( Site 0038), Baltimore, Maryland
  - Henry Ford Hospital ( Site 0024), Detroit, Michigan
  - St. Vincent Frontier Cancer Center ( Site 0005), Billings, Montana
  - Providence Portland Medical Center ( Site 0019), Portland, Oregon
  - Thomas Jefferson University - Clinical Trials Office ( Site 0027), Philadelphia, Pennsylvania
  - Inova Schar Cancer Institute ( Site 0022), Fairfax, Virginia
  - Blue Ridge Cancer Care ( Site 0036), Roanoke, Virginia
  - Northwest Medical Specialties, PLLC ( Site 0033), Tacoma, Washington
- Argentina (5):
  - Hospital Británico de Buenos Aires-Oncology ( Site 0308), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Fundación favaloro para la Docencia e Investigación Médica-Oncología ( Site 0301), Buenos Aires, Buenos Aires F.D.
  - Instituto de Oncología de Rosario ( Site 0305), Rosario, Santa Fe Province
  - Centro de Educación Médica e Investigaciones Clínicas (CEMIC)-Medical Oncology ( Site 0303), Buenos Aires
  - IDIM - Instituto de Diagnóstico e Investigaciones Metabólicas ( Site 0300), Buenos Aires
- Australia (6):
  - Royal Brisbane and Women's Hospital-Medical Oncology Clinical Trials Unit, Cancer Care Services ( Si, Brisbane, Queensland
  - Gallipoli Medical Research Foundation-GMRF CTU ( Site 1500), Greenslopes, Queensland
  - The Queen Elizabeth Hospital-Cancer Clinical Trials ( Site 1503), Woodville, South Australia
  - Epworth Freemasons ( Site 1506), Melbourne, Victoria
  - Western Health-Sunshine & Footscray Hospitals ( Site 1501), St Albans, Victoria
  - Hollywood Private Hospital-Medical Oncology ( Site 1507), Perth, Western Australia
- Canada (6):
  - Cross Cancer Institute-Department of Medical Oncology ( Site 0207), Edmonton, Alberta
  - NSHA-QEII Health Sciences Centre-Dickson Bldg-Dept. of Medical Oncology ( Site 0200), Halifax, Nova Scotia
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0205), Hamilton, Ontario
  - North York General Hospital ( Site 0206), Toronto, Ontario
  - CIUSSS de l'Est-de-l'Île-de-Montréal ( Site 0211), Montreal, Quebec
  - CHU de Quebec - Université Laval - Hotel Dieu de Quebec-Hemato-Dermato-Gyneco-Oncology ( Site 0203), Québec, Quebec
- China (3):
  - The First People's Hospital of Foshan-Gastrointestinal oncology ( Site 1604), Foshan, Guangdong
  - SUN YAT-SEN UNIVERSITY CANCER CENTRE ( Site 1600), Guangzhou, Guangdong
  - Sir Run Run Shaw Hospital-Medical Oncology ( Site 1606), Hangzhou, Zhejiang
- Denmark (4):
  - Rigshospitalet ( Site 0702), Copenhagen, Capital Region
  - Herlev and Gentofte Hospital-Department of Oncology ( Site 0704), Copenhagen, Capital Region
  - Odense Universitetshospital ( Site 0700), Odense, Region Syddanmark
  - Vejle Sygehus-Department of Oncology ( Site 0701), Vejle, Region Syddanmark
- Germany (5):
  - Klinikum am Steinenberg-Kreiskliniken Reutlingen GmbH ( Site 0908), Reutlingen, Baden-Wurttemberg
  - klinikum rechts der isar der technischen universität münchen-Klinik und Poliklinik für Innere Mediz, Munich, Bavaria
  - Onkodok GmbH ( Site 0907), Gütersloh, North Rhine-Westphalia
  - Charité Universitaetsmedizin Berlin - Campus Mitte ( Site 0901), Berlin
  - Asklepios Altona-Oncology ( Site 0903), Hamburg
- Israel (5):
  - Rambam Health Care Campus-Oncology ( Site 0800), Haifa
  - Shaare Zedek Medical Center-Oncology ( Site 0804), Jerusalem
  - Hadassah Medical Center-Oncology ( Site 0802), Jerusalem
  - Sheba Medical Center ( Site 0803), Ramat Gan
  - Sourasky Medical Center-Oncology ( Site 0801), Tel Aviv
- Japan (11):
  - Aichi Cancer Center Hospital ( Site 1701), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 1700), Kashiwa, Chiba
  - Kobe City Medical Center General Hospital ( Site 1707), Kobe, Hyōgo
  - Kagawa University Hospital ( Site 1708), Kita, Kagawa-ken
  - Kanagawa cancer center ( Site 1705), Yokohama, Kanagawa
  - Kindai University Hospital- Osakasayama Campus-Medical Oncology ( Site 1704), Sayama, Osaka
  - Saitama Prefectural Cancer Center ( Site 1703), Ina-machi, Saitama
  - Shizuoka Cancer Center ( Site 1706), Nakatogari, Shizuoka
  - National Hospital Organization Kyushu Cancer Center ( Site 1709), Fukuoka
  - National Cancer Center Hospital ( Site 1702), Tokyo
  - Japanese Foundation for Cancer Research-GI Oncology ( Site 1710), Tokyo
- Russia (7):
  - GBUZ Republican Clinical Oncological Dispensary-Antitumor drug therapy department ( Site 1109), Ufa, Baskortostan, Respublika
  - Saint-Petersburg City Clinical Oncology Dispensary-Department of chemotherapy ( Site 1100), Saint Petersburg, Leningradskaya Oblast'
  - The National Medico-Surgical Center N.I. Pirogov ( Site 1102), Moscow, Moscow
  - Fed State Budgetary Inst N.N. Blokhin Med Center of Oncology MHRF ( Site 1107), Moscow, Moscow
  - First Moscow State Medical University I.M. Sechenov-Interhospital Institution ""Health Management (, Moscow, Moscow
  - SVERDLOVSK REGIONAL ONCOLOGY DISPENSARY ( Site 1108), Yekaterinburg, Sverdlovsk Oblast
  - SHBI Leningrad Regional Clinical Oncology Dispensary-Clinical Trials Department ( Site 1111), Saint Petersburg
- South Korea (6):
  - Korea University Anam Hospital ( Site 1806), Seoul
  - Seoul National University Hospital-Internal Medicine ( Site 1800), Seoul
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 1801), Seoul
  - Asan Medical Center ( Site 1803), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 1804), Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital ( Site 1802), Seoul
- Spain (5):
  - Hospital Universitario Marqués de Valdecilla ( Site 1201), Santander, Cantabria
  - Hospital Universitario Central de Asturias-Digestive ( Site 1200), Oviedo, Principality of Asturias
  - Hospital Universitari Vall d'Hebron-Oncology ( Site 1204), Barcelona
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON ( Site 1205), Madrid
  - Hospital Universitario Virgen de Valme-Departamento de Oncologia ( Site 1207), Seville
- Taiwan (5):
  - China Medical University Hospital-Surgical Department ( Site 1903), Taichung
  - NATIONAL CHENG-KUNG UNI. HOSP. ( Site 1904), Tainan
  - National Taiwan University Hospital ( Site 1900), Taipei
  - Taipei Veterans General Hospital-Oncology ( Site 1901), Taipei
  - Chang Gung Medical Foundation.Linkou Branch ( Site 1902), Taoyuan District
- Turkey (Türkiye) (8):
  - Hacettepe Universitesi-oncology hospital ( Site 1302), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 1304), Ankara
  - Trakya University-Oncology ( Site 1303), Edirne
  - Acıbadem Maslak Hastanesi ( Site 1307), Istanbul
  - Istanbul Universitesi Cerrahpasa-Medical Oncology ( Site 1300), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 1301), Istanbul
  - Ege University Medicine of Faculty-Medical Oncology ( Site 1305), Izmir
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi ( Site 1306), Malatya
- United Kingdom (7):
  - Addenbrooke's Hospital ( Site 1407), Cambridge, Cambridgeshire
  - UCLH-Cancer Clinical Trials Unit ( Site 1400), London, Essex
  - Guy's & St Thomas' NHS Foundation Trust ( Site 1404), London, London, City of
  - ROYAL MARSDEN HOSPITAL (CHELSEA) ( Site 1403), London, London, City of
  - Western General Hospital ( Site 1401), Edinburgh, Midlothian
  - Royal Marsden Hospital (Sutton) ( Site 1409), London, Surrey
  - The Christie-Medical Oncology ( Site 1411), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Kawazoe A, Xu RH, Garcia-Alfonso P, Passhak M, Teng HW, Shergill A, Gumus M, Qvortrup C, Stintzing S, Towns K, Kim TW, Shiu KK, Cundom J, Ananda S, Lebedinets A, Fu R, Jain R, Adelberg D, Heinemann V, Yoshino T, Elez E; LEAP-017 Investigators. Lenvatinib Plus Pembrolizumab Versus Standard of Care for Previously Treated Metastatic Colorectal Cancer: Final Analysis of the Randomized, Open-Label, Phase III LEAP-017 Study. J Clin Oncol. 2024 Aug 20;42(24):2918-2927. doi: 10.1200/JCO.23.02736. Epub 2024 Jun 4. PMID 38833658
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26865&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 480 participants were enrolled in the Global Cohort, including 17 participants from China. An additional 83 participants were subsequently enrolled in the China extension, bringing the total number of participants in the China Cohort to 100 and the overall study population to 563. These results have been updated to include data from the China Cohort.
Pre-assignment Details: Primary Completion for the study is being updated to 27-Sep-2024 to reflect that the protocol specified non-alpha controlled final analyses for the China Cohort was conducted with a 27-Sep 2024 data cutoff, after the protocol-specified final analyses of the Global Cohort was completed on 20-Feb-2023. Final Analysis of all outcome measures for the Global Cohort was conducted with a data cut-off of 20-Feb-2023.
Groups:
- Lenvatinib+Pembrolizumab: Participants received pembrolizumab 400 mg via intravenous (IV) infusion on Day 1 of each 6-week (Q6W) Cycle for up to 18 cycles (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule once daily until progressive disease.
- Standard of Care (SOC) Treatment: Participants received regorafenib 160 mg via oral tablet once daily on Days 1 through 21 of each 4-week cycle OR TAS-102 (trifluridine and tipiracil hydrochloride) 35 mg/m^2 via oral tablet twice a day on Days 1 through 5 and Days 8-12 of each 4-week cycle until progressive disease.
Period: Overall Study
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Started | 282 | 281
Treated | 279 | 277
Global Cohort Efficacy | 241 | 239
China Cohort Efficacy | 53 (Includes 12 participants who were also enrolled in the Global Cohort) | 47 (Includes 5 participants who were also enrolled in the Global Cohort)
Global Cohort Safety | 238 | 235
China Cohort Safety | 53 (Includes 12 participants who were also enrolled in the Global Cohort) | 47 (Includes 5 participants who were also enrolled in the Global Cohort)
Completed | 0 | 0
Not Completed | 282 | 281
Not completed — Death | 249 | 260
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Parent/Guardian | 0 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Sponsor Decision | 30 | 15

BASELINE CHARACTERISTICS:
Population: Baseline characteristics include data from 480 participants in the Global Cohort and 83 participants from the China extension (Total Study N=563)
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment | Total
Number analyzed (Participants) | 282 | 281 | 563
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.1 (11.7) | 57.2 (11.7) | 57.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 116 | 237
  Male | 161 | 165 | 326
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 13 | 39
  Not Hispanic or Latino | 255 | 267 | 522
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 122 | 123 | 245
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 152 | 152 | 304
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 2 | 4
Presence of Liver Metastasis [Count of Participants; unit: Participants] — Number of participants with liver metastasis at baseline (Yes/No)
  Participants
    Yes | 192 | 190 | 382
    No | 90 | 91 | 181

OUTCOME MEASURES:

1. Secondary Outcome: Global Cohort: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from date of randomization to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. PFS as assessed by BICR per modified RECIST 1.1 is presented. Per the sSAP, Final Analysis for the Global Cohort was performed with a data cut-off date of 20-Feb-2023.
Time Frame: Up to approximately 22 months (through sSAP pre-specified Final Analysis database cut-off date of 20-Feb-2023)
Population: All randomized participants in the Global Cohort included in the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 241 | 239
Months | 3.8 [3.7 to 5.1] | 3.3 [2.0 to 3.7]
Statistical Analysis 1: Comparison: Lenvatinib+Pembrolizumab vs Standard of Care (SOC) Treatment; Test type: Other — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by presence of liver metastasis (Yes/No); p = 0.0003, Log Rank — One-sided p-value based on log-rank test stratified by presence of liver metastasis; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.56 to 0.85]

2. Secondary Outcome: China Cohort: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from date of randomization to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. PFS as assessed by BICR per modified RECIST 1.1 is presented. Per the sSAP, the China Cohort was evaluated for efficacy separately from the Global Cohort, with Final Analysis performed using a data cut-off of 27-Sep-2024.
Time Frame: Up to approximately 35 months (through sSAP pre-specified Final Analysis database cut-off date of 27-Sep-2024)
Population: All randomized participants in the China Cohort (17 participants enrolled in the Global Cohort and 83 participants enrolled in the China extension) included in the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Lenvatinib+Pembrolizumab: Participants enrolled in China received pembrolizumab 400 mg via intravenous (IV) infusion on Day 1 of each 6-week (Q6W) Cycle for up to 18 cycles (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule once daily until progressive disease.
- Standard of Care (SOC) Treatment: Participants enrolled in China received regorafenib 160 mg via oral tablet once daily on Days 1 through 21 of each 4-week cycle OR TAS-102 (trifluridine and tipiracil hydrochloride) 35 mg/m^2 via oral tablet twice a day on Days 1 through 5 and Days 8-12 of each 4-week cycle until progressive disease.
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 53 | 47
Months | 3.7 [2.9 to 3.9] | 2.4 [1.9 to 5.4]
Statistical Analysis 1: Comparison: Lenvatinib+Pembrolizumab vs Standard of Care (SOC) Treatment; Test type: Other — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; p = 0.7421, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 1.15, 85% CI 2-sided [0.75 to 1.77]

3. Secondary Outcome: Global Cohort: Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by BICR
Description: ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. ORR per modified RECIST 1.1 assessed by BICR is presented. Per the sSAP, Final Analysis for the Global Cohort was performed with a data cut-off date of 20-Feb-2023.
Time Frame: Up to approximately 22 months (through sSAP pre-specified Final Analysis database cut-off date of 20-Feb-2023)
Population: All randomized participants in the Global Cohort included in the treatment arm to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 241 | 239
Percentage of Participants | 10.4 [6.8 to 14.9] | 1.7 [0.5 to 4.2]
Statistical Analysis 1: Comparison: Lenvatinib+Pembrolizumab vs Standard of Care (SOC) Treatment; Test type: Other; p < 0.0001, Chi-squared; Difference in Percentage vs. SOC = 8.7, 95% CI 2-sided [4.7 to 13.5] — Based on Miettinen & Nurminen method stratified by presence of liver metastasis

4. Secondary Outcome: China Cohort: Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by BICR
Description: ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. ORR per modified RECIST 1.1 assessed by BICR is presented. Per the sSAP, the China Cohort was evaluated for efficacy separately from the Global Cohort, with Final Analysis performed using a data cut-off of 27-Sep-2024.
Time Frame: Up to approximately 35 months (through sSAP pre-specified Final Analysis database cut-off date of 27-Sep-2024)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 53 | 47
Percentage of Participants | 7.5 [2.1 to 18.2] | 4.3 [0.5 to 14.5]
Statistical Analysis 1: Comparison: Lenvatinib+Pembrolizumab vs Standard of Care (SOC) Treatment; Test type: Other; p = 0.2456, Chi-squared; Difference in Percentage vs. SOC = 3.3, 95% CI 2-sided [-7.7 to 14.3] — Based on Miettinen & Nurminen method

5. Secondary Outcome: Global Cohort: Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR
Description: For participants who demonstrated CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions), DOR is defined as the time from the first documented evidence of CR or PR until PD or death from any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, or death from any cause, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR per modified RECIST 1.1 is presented. Per the sSAP, Final Analysis for the Global Cohort was performed with a data cut-off date of 20-Feb-2023.
Time Frame: Up to approximately 22 months (through sSAP pre-specified Final Analysis database cut-off date of 20-Feb-2023)
Population: Randomized participants in the Global Cohort who had a confirmed complete or partial response, included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 25 | 4
Months | 11.1 [7.7 to NA] — NA=Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse | 7.6 [6.0 to NA] — NA=Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse

6. Secondary Outcome: China Cohort: Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR
Description: For participants who demonstrated CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions), DOR is defined as the time from the first documented evidence of CR or PR until PD or death from any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, or death from any cause, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR per modified RECIST 1.1 is presented. Per the sSAP, the China Cohort was evaluated for efficacy separately from the Global Cohort, with Final Analysis performed using a data cut-off of 27-Sep-2024.
Time Frame: Up to approximately 35 months (through sSAP pre-specified Final Analysis database cut-off date of 27-Sep-2024)
Population: Randomized participants in the China Cohort (17 participants enrolled in the Global Cohort and 83 participants enrolled in the China extension) who had a confirmed complete or partial response, included in the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 4 | 2
Months | 4.4 [3.5 to NA] — NA=Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse | NA [9.1 to NA] — NA=Median duration and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse

7. Secondary Outcome: Global Cohort: Number of Participants Who Experience an Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Per the sSAP, Final Analysis for the Global Cohort was performed with a data cut-off date of 20-Feb-2023.
Time Frame: Up to approximately 22 months (through sSAP pre-specified Final Analysis database cut-off date of 20-Feb-2023)
Population: All randomized participants in the Global Cohort who received at least one dose of study treatment. Two participants randomized to pembrolizumab plus lenvatinib group were incorrectly treated with SOC; these participants were included in the SOC group for safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 238 | 235
Participants | 237 | 230

8. Secondary Outcome: China Cohort: Number of Participants Who Experience an Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Per the sSAP, the China Cohort was evaluated for safety separately from the Global Cohort, with Final Analysis performed using a data cut-off of 27-Sep-2024.
Time Frame: Up to approximately 35 months (through sSAP pre-specified Final Analysis database cut-off date of 27-Sep-2024)
Population: All randomized participants in the China Cohort (17 participants enrolled in the Global Cohort and 83 participants enrolled in the China extension) who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 53 | 47
Participants | 53 | 47

9. Secondary Outcome: Global Cohort: Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued any study treatment due to an adverse event is presented. Per the sSAP, Final Analysis for the Global Cohort was performed with a data cut-off date of 20-Feb-2023.
Time Frame: Up to approximately 22 months (through sSAP pre-specified Final Analysis database cut-off date of 20-Feb-2023)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 238 | 235
Participants | 37 | 10

10. Secondary Outcome: China Cohort: Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued any study treatment due to an adverse event is presented. Per the sSAP, the China Cohort was evaluated for safety separately from the Global Cohort, with Final Analysis performed using a data cut-off of 27-Sep-2024.
Time Frame: Up to approximately 28 months (through sSAP pre-specified Final Analysis database cut-off date of 27-Sep-2024)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 53 | 47
Participants | 8 | 5

11. Secondary Outcome: Global Cohort: Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score
Description: The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to the questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and Quality of Life (QoL; "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in GHS (EORTC QLQ-C30 Item 29) and QoL (EORTC QLQ-C30 Item 30) combined score is presented. A higher score indicates a better outcome.
Time Frame: Baseline and 8 weeks
Population: All participants in the Global Cohort who have at least one assessment available for EORTC QLQ-C30 and have received at least one dose of the study intervention. Per the sSAP, this Patient Reported Outcome (PRO) was not pre-specified for the China Cohort and was thus not analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 234 | 229
Scores on a scale | -4.91 [-7.67 to -2.14] | -7.62 [-10.48 to -4.76]
Statistical Analysis 1: Comparison: Lenvatinib+Pembrolizumab vs Standard of Care (SOC) Treatment; Test type: Other; p = 0.1553, cLDA model — Based on a cLDA model with the PRO scores as the response variable with covariates for treatment by study visit interaction and stratification factor presence of liver metastasis (Yes/No); Difference in least squares means = 2.71, 95% CI 2-sided [-1.03 to 6.46]

12. Secondary Outcome: Global Cohort: Change From Baseline in EORTC QLQ-C30 Physical Functioning (Items 1-5) Score
Description: The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 5 questions about their physical functioning (Items 1-5) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores meant a better level of function. The change from baseline in the EORTC QLQ-C30 Physical Functioning (Items 1-5) scale score is presented.
Time Frame: Baseline and 8 weeks
Population: All participants in the Global Cohort who have at least one assessment available for EORTC QLQ-C30 and have received at least one dose of the study intervention. Per the sSAP, this PRO was not pre-specified for the China Cohort and was thus not analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 234 | 229
Scores on a scale | -6.16 [-8.51 to -3.82] | -7.32 [-9.75 to -4.90]
Statistical Analysis 1: Comparison: Lenvatinib+Pembrolizumab vs Standard of Care (SOC) Treatment; Test type: Other; p = 0.4967, cLDA model — [p-value comment as in outcome 11, analysis 1]; Difference in LS means = 1.16, 95% CI 2-sided [-2.19 to 4.51]

13. Secondary Outcome: Global Cohort: Change From Baseline in EORTC QLQ-C30 Appetite Loss (Item 13) Score
Description: The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire, including a single-item scale score for appetite loss (QLQ-C30 Item 13). For this item, individual responses to the question "Have you lacked appetite?" are given on a 4-point scale (1=Not at all; 4=Very much). Scores are transformed to a range from 0-100, with a lower score indicating a better outcome. The change from baseline in the EORTC QLQ-C30 appetite loss (Item 13) scale score is presented.
Time Frame: Baseline and 8 weeks
Population: All participants in the Global Cohort who have at least one assessment available for EORTC QLQ-C30 appetite loss and have received at least one dose of the study intervention. Per the sSAP, this PRO was not pre-specified for the China Cohort and was thus not analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 234 | 230
Scores on a scale | 12.44 [8.50 to 16.38] | 9.08 [5.00 to 13.15]
Statistical Analysis 1: Comparison: Lenvatinib+Pembrolizumab vs Standard of Care (SOC) Treatment; Test type: Other; p = 0.2271, cLDA model — [p-value comment as in outcome 11, analysis 1]; Difference in LS means = 3.36, 95% CI 2-sided [-2.10 to 8.82]

14. Secondary Outcome: Global Cohort: Change From Baseline in EORTC Quality of Life Questionnaire-Colorectal Cancer-Specific 29 Items (QLQ-CR29) Bloating (Item 37) Score
Description: The EORTC QLQ-CR29 is a health-related quality-of life (QoL) questionnaire specific for colorectal cancer, including a single-item scale score for bloating (QLQ-CR29 Item 37). For this item, individual responses to the question "Did you have a bloated feeling in your abdomen?" are given on a 4-point scale (1=Not at all; 4=Very much). Scores are transformed to a range from 0-100, with a lower score indicating a better outcome. The change from baseline in the EORTC QLQ-CR29 bloating (Item 37) scale score is presented.
Time Frame: Baseline and 8 weeks
Population: All participants in the Global Cohort who have at least one assessment available for EORTC QLQ-CR29 and have received at least one dose of the study intervention. Per the sSAP, this PRO was not pre-specified for the China Cohort and was thus not analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 234 | 230
Scores on a scale | -0.30 [-3.78 to 3.19] | 5.16 [1.56 to 8.77]
Statistical Analysis 1: Comparison: Lenvatinib+Pembrolizumab vs Standard of Care (SOC) Treatment; Test type: Other; p = 0.0264, cLDA model — [p-value comment as in outcome 11, analysis 1]; Difference in LS means = -5.46, 95% CI 2-sided [-10.27 to -0.65]

15. Secondary Outcome: Global Cohort: Time to Deterioration (TTD) in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score
Description: TTD is defined as the time from baseline to the first onset of a ≥10-point deterioration (decrease) from baseline in Global Health Status (GHS; EORTC QLQ-C30 Item 29) & Quality of Life (QoL; EORTC QLQ-C30 Item 30) combined score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from baseline in GHS and QoL combined score, is presented. A longer TTD indicates a better outcome.
Time Frame: Up to approximately 21 months
Population: All participants in the Global Cohort who have at least one assessment available for EORTC QLQ-C30 GHS/QoL TTD and have received at least one dose of the study intervention. Per the sSAP, this PRO was not pre-specified for the China Cohort and was thus not analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 227 | 220
Months | 1.4 [1.1 to 1.9] | 1.4 [1.0 to 1.8]
Statistical Analysis 1: Comparison: Lenvatinib+Pembrolizumab vs Standard of Care (SOC) Treatment; Test type: Other; p = 0.4338, Regression, Cox; Two-sided p-value based on log-rank test stratified by presence of liver metastasis (Yes/No); Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.73 to 1.14]

16. Secondary Outcome: Global Cohort: TTD in EORTC QLQ-C30 Physical Functioning (Items 1-5) Score
Description: TTD is defined as the time from baseline to the first onset of a ≥10-point deterioration (decrease) from baseline in physical functioning score (QLQ-C30 Items 1-5). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from baseline in physical functioning score, is presented. A longer TTD indicates a better outcome.
Time Frame: Up to approximately 21 months
Population: All participants in the Global Cohort who have at least one assessment available for EORTC QLQ-C30 Physical Functioning TTD and have received at least one dose of the study intervention. Per the sSAP, this PRO was not pre-specified for the China Cohort and was thus not analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 226 | 221
Months | 1.8 [1.4 to 2.0] | 2.0 [1.4 to 2.3]
Statistical Analysis 1: Comparison: Lenvatinib+Pembrolizumab vs Standard of Care (SOC) Treatment; Test type: Other; p = 0.4316, Regression, Cox — Two-sided p-value based on log-rank test stratified by presence of liver metastasis (Yes/No); Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.87 to 1.38]

17. Secondary Outcome: Global Cohort: TTD in EORTC QLQ-C30 Appetite Loss (Item 13) Score
Description: TTD is defined as the time from baseline to the first onset of a ≥10-point deterioration (increase) from baseline in appetite loss (QLQ-C30 Item 13) score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point change (increase) from baseline in appetite loss score, is presented. A longer TTD indicates a better outcome.
Time Frame: Up to approximately 21 months
Population: All participants in the Global Cohort who have at least one assessment available for EORTC QLQ-C30 Appetite Loss TTD and have received at least one dose of the study intervention. Per the sSAP, this PRO was not pre-specified for the China Cohort and was thus not analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 226 | 221
Months | 1.4 [1.1 to 1.8] | 1.4 [1.1 to 1.9]
Statistical Analysis 1: Comparison: Lenvatinib+Pembrolizumab vs Standard of Care (SOC) Treatment; Test type: Other; p = 0.5587, Regression, Cox; Two-sided p-value based on log-rank test stratified by presence of liver metastasis (Yes/No); Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.85 to 1.32]

18. Secondary Outcome: Global Cohort: TTD in EORTC Quality of Life Questionnaire-Colorectal Cancer-Specific 29 Items (QLQ-CR29) Bloating (Item 37) Score
Description: TTD is defined as the time from baseline to the first onset of a ≥10-point deterioration (increase) from baseline in bloating (QLQ-CR29 Item 37) score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point change (increase) from baseline in bloating score, is presented. A longer TTD indicates a better outcome.
Time Frame: Up to approximately 21 months
Population: All participants in the Global Cohort who have at least one assessment available for EORTC QLQ-CR29 Bloating TTD and have received at least one dose of the study intervention. Per the sSAP, this PRO was not pre-specified for the China Cohort and was thus not analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 224 | 221
Months | 3.4 [2.3 to 5.2] | 3.2 [2.3 to 5.6]
Statistical Analysis 1: Comparison: Lenvatinib+Pembrolizumab vs Standard of Care (SOC) Treatment; Test type: Other; p = 0.6794, Regression, Cox — Two-sided p-value based on log-rank test stratified by presence of liver metastasis (Yes/No); Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.73 to 1.23]

19. Primary Outcome: Global Cohort: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death from any cause. Per the supplemental Statistical Analysis Plan (sSAP), Final Analysis for the Global Cohort was performed with a data cut-off date of 20-Feb-2023.
Time Frame: Up to approximately 22 months (through sSAP pre-specified Final Analysis database cut-off date of 20-Feb-2023)
Population: All randomized participants in the Global Cohort included in the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 241 | 239
Months | 9.8 [8.4 to 11.6] | 9.3 [8.2 to 10.9]
Statistical Analysis 1: Comparison: Lenvatinib+Pembrolizumab vs Standard of Care (SOC) Treatment; Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by presence of liver metastasis (Yes/No); Test type: Superiority; p = 0.0379, Log Rank; One-sided p-value based on log-rank test stratified by presence of liver metastasis (Yes/No); Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.68 to 1.02] — HR=Lenvatinib + pembrolizumab vs. SOC treatment

20. Primary Outcome: China Cohort: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death from any cause. Per the sSAP, the China Cohort was evaluated for efficacy separately from the Global Cohort, with Final Analysis performed using a data cut-off of 27-Sep-2024.
Time Frame: Up to approximately 35 months (through sSAP pre-specified Final Analysis database cut-off date of 27-Sep-2024)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib+Pembrolizumab | Standard of Care (SOC) Treatment
Number analyzed (Participants) | 53 | 47
Months | 10.9 [8.8 to 16.5] | 10.2 [6.1 to 12.7]
Statistical Analysis 1: Comparison: Lenvatinib+Pembrolizumab vs Standard of Care (SOC) Treatment; Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Test type: Superiority; p = 0.3574, Log Rank; One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.60 to 1.42] — HR=Lenvatinib + pembrolizumab vs. SOC treatment

ADVERSE EVENTS:
Time Frame: Up to approximately 41 months (through End of Trial database cut-off date of 27-Sep-2024)
Description: The population for all-cause mortality includes all participants (N=563) in the treatment arm to which they were randomized. Serious and other AEs include all treated participants according to treatment received. 2 participants randomized to lenvatinib plus pembrolizumab were incorrectly treated with SOC and were included in SOC arm. Per protocol, MedDRA V27.0 terms 'Neoplasm progression' 'Malignant neoplasm progression' and 'Disease progression' not related to the drug are excluded.
Groups:
- Lenvatinib + Pembrolizumab: Participants received pembrolizumab 400 mg via intravenous (IV) infusion on Day 1 of each 6-week (Q6W) Cycle for up to 18 cycles (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule once daily until progressive disease.
- Standard Of Care Treatment: Participants received regorafenib 160 mg via oral tablet once daily on Days 1 through 21 of each 4-week cycle OR TAS-102 (trifluridine and tipiracil hydrochloride) 35 mg/m^2 via oral tablet twice a day on Days 1 through 5 and Days 8-12 of each 4-week cycle until progressive disease.
Arm/Group | Lenvatinib + Pembrolizumab | Standard Of Care Treatment
All-Cause Mortality (participants affected / at risk) | 251/282 | 264/281
Serious Adverse Events (participants affected / at risk) | 117/279 | 66/277
Other Adverse Events (participants affected / at risk) | 273/279 | 263/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab (N=279) | Standard Of Care Treatment (N=277)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 6 (6)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (4)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 5 (5) | 3 (3)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immune-mediated pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Asthenia (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 4 (4)
Biliary obstruction (Hepatobiliary disorders) | 2 (2) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 1 (2) | 3 (4)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (3) | 0 (0)
Malignant biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Fournier's gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (2)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (4) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Spontaneous bacterial peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (7) | 4 (5)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma prolapse (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (3) | 1 (1)
Clostridium test positive (Investigations) | 1 (1) | 0 (0)
Granulocyte count decreased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (5) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Immune-mediated nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic fluid collection (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 6 (6) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab (N=279) | Standard Of Care Treatment (N=277)
Anaemia (Blood and lymphatic system disorders) | 49 (64) | 60 (73)
Neutropenia (Blood and lymphatic system disorders) | 8 (22) | 33 (82)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (25) | 12 (18)
Hyperthyroidism (Endocrine disorders) | 14 (15) | 4 (5)
Hypothyroidism (Endocrine disorders) | 105 (112) | 19 (23)
Abdominal distension (Gastrointestinal disorders) | 16 (21) | 14 (15)
Abdominal pain (Gastrointestinal disorders) | 58 (69) | 45 (56)
Abdominal pain upper (Gastrointestinal disorders) | 27 (29) | 16 (20)
Constipation (Gastrointestinal disorders) | 43 (51) | 44 (58)
Diarrhoea (Gastrointestinal disorders) | 119 (231) | 64 (85)
Dry mouth (Gastrointestinal disorders) | 24 (27) | 20 (21)
Nausea (Gastrointestinal disorders) | 66 (77) | 87 (139)
Stomatitis (Gastrointestinal disorders) | 30 (31) | 16 (18)
Vomiting (Gastrointestinal disorders) | 60 (83) | 49 (84)
Asthenia (General disorders) | 49 (62) | 36 (45)
Fatigue (General disorders) | 78 (88) | 67 (81)
Malaise (General disorders) | 14 (15) | 16 (18)
Mucosal inflammation (General disorders) | 18 (20) | 8 (8)
Oedema peripheral (General disorders) | 26 (26) | 8 (8)
Pyrexia (General disorders) | 40 (50) | 24 (32)
COVID-19 (Infections and infestations) | 27 (29) | 12 (12)
Urinary tract infection (Infections and infestations) | 28 (39) | 15 (17)
Alanine aminotransferase increased (Investigations) | 50 (68) | 30 (38)
Amylase increased (Investigations) | 16 (17) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 67 (90) | 39 (49)
Blood alkaline phosphatase increased (Investigations) | 27 (33) | 17 (17)
Blood bilirubin increased (Investigations) | 46 (60) | 41 (52)
Blood creatinine increased (Investigations) | 21 (30) | 8 (11)
Blood thyroid stimulating hormone increased (Investigations) | 37 (57) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 14 (15) | 9 (9)
Neutrophil count decreased (Investigations) | 14 (34) | 48 (151)
Platelet count decreased (Investigations) | 60 (91) | 32 (59)
Weight decreased (Investigations) | 65 (69) | 26 (27)
White blood cell count decreased (Investigations) | 15 (20) | 36 (118)
Decreased appetite (Metabolism and nutrition disorders) | 75 (90) | 69 (95)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 34 (43) | 13 (18)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (23) | 18 (25)
Hyponatraemia (Metabolism and nutrition disorders) | 19 (23) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 50 (66) | 17 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 34 (37) | 26 (29)
Myalgia (Musculoskeletal and connective tissue disorders) | 29 (30) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (22) | 10 (10)
Dizziness (Nervous system disorders) | 19 (19) | 21 (24)
Headache (Nervous system disorders) | 45 (61) | 14 (17)
Insomnia (Psychiatric disorders) | 19 (21) | 20 (20)
Proteinuria (Renal and urinary disorders) | 136 (200) | 42 (63)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (39) | 24 (27)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 57 (62) | 21 (24)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 21 (24)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 59 (78) | 60 (74)
Pruritus (Skin and subcutaneous tissue disorders) | 20 (23) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 39 (44) | 17 (17)
Hypertension (Vascular disorders) | 156 (221) | 63 (81)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT04776148/Prot_001.pdf
  • Statistical Analysis Plan (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT04776148/SAP_002.pdf